CLINICAL TRIAL: NCT03010631
Title: Comparative Pharmacokinetics and Food-Effect Bioavailability of a Sprinkle Formulation of Lubiprostone After Oral Administration in Healthy Volunteers
Brief Title: Comparative Pharmacokinetics and Food-Effect Bioavailability of Lubiprostone Sprinkle in Healthy Volunteers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sucampo Pharma Americas, LLC (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SCMP-0211-304
Record Dates: First submitted 2016-12-20; First posted 2017-01-05 (Estimated); Results first posted 2020-03-09 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2018-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Lubiprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Treatment Sequence AB) (Active Comparator): Cohort 1: Treatment A. Capsule Fasted (7-day Washout) then Treatment B. Sprinkle Formulation, Fasted
  Interventions: Drug: Cohort 1: Lubiprostone Capsule, Fasted; Drug: Cohort 1: Lubiprostone Sprinkle Formulation, Fasted
- Cohort 1 (Treatment Sequence BA) (Experimental): Cohort 1: Treatment B. Sprinkle Formulation, Fasted (7-day Washout) then Treatment A. Capsule Fasted
  Interventions: Drug: Cohort 1: Lubiprostone Capsule, Fasted; Drug: Cohort 1: Lubiprostone Sprinkle Formulation, Fasted
- Cohort 2 (Treatment Sequence CD) (Experimental): Cohort 2: Treatment C: Sprinkle Formulation, Fed (7-day Washout) then Treatment D: Sprinkle Formulation, Fasted
  Interventions: Drug: Cohort 2: Lubiprostone Sprinkle Formulation, Fed; Drug: Cohort 2: Lubiprostone Sprinkle Formulation, Fasted
- Cohort 2 (Treatment Sequence DC) (Experimental): Cohort 2: Treatment D: Sprinkle Formulation, Fasted (7-day Washout) then Treatment C. Sprinkle Formulation, Fed
  Interventions: Drug: Cohort 2: Lubiprostone Sprinkle Formulation, Fed; Drug: Cohort 2: Lubiprostone Sprinkle Formulation, Fasted

INTERVENTIONS:
Drug: Cohort 1: Lubiprostone Capsule, Fasted — Lubiprostone soft gelatin capsule administered under fasted conditions
  Other Names: AMITIZA®; Treatment A
  Arms: Cohort 1 (Treatment Sequence AB); Cohort 1 (Treatment Sequence BA)
Drug: Cohort 1: Lubiprostone Sprinkle Formulation, Fasted — Lubiprostone sprinkle formulation administered under fasted conditions
  Other Names: Lubiprostone microbeads; Treatment B
  Arms: Cohort 1 (Treatment Sequence AB); Cohort 1 (Treatment Sequence BA)
Drug: Cohort 2: Lubiprostone Sprinkle Formulation, Fed — Lubiprostone sprinkle formulation administered under fed conditions
  Other Names: Lubiprostone microbeads; Treatment C
  Arms: Cohort 2 (Treatment Sequence CD); Cohort 2 (Treatment Sequence DC)
Drug: Cohort 2: Lubiprostone Sprinkle Formulation, Fasted — Lubiprostone sprinkle formulation administered under fasted conditions
  Other Names: Lubiprostone microbeads; Treatment D
  Arms: Cohort 2 (Treatment Sequence CD); Cohort 2 (Treatment Sequence DC)

SUMMARY:
A study to compare the pharmacokinetics and food-effect bioavailability of sprinkle formulation of lubiprostone, as compared to lubiprostone capsules in healthy volunteers.

DETAILED DESCRIPTION:
To compare the pharmacokinetics of the sprinkle formulation of lubiprostone, as compared to lubiprostone capsules and to determine the effect of food on the bioavailability and plasma pharmacokinetics of lubiprostone sprinkle.

ELIGIBILITY:
Inclusion Criteria:

* Is male or female, between 18 and 55 years of age, inclusive.
* Has a 12-lead electrocardiogram (ECG) within normal limits and is in good health based upon review of medical history, physical examination results, vital signs (within normal range), and normal laboratory profile for both blood and urine.

Exclusion Criteria:

* Has an active or recent history of alcoholism or drug addiction (within 1 year prior)
* Is a smoker or has a recent history of smoking (within 6 months)
* Routinely consumes food known to alter drug metabolism (i.e., grapefruit juice, coffee, tea, cola, chocolate, cocoa, or other caffeine or methyl-xanthine containing foods or beverages) and/or cannot refrain from these items
* Has donated blood within 3 months
* Has a medical/surgical condition that might interfere with the absorption, distribution, metabolism, or excretion of the study medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2016-11-16 (Actual); Primary Completion 2016-12-23 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Mallinckrodt
Locations (1):
- ICON, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adams A, Barish C, Chen A, Dennis P, Krause R, Lichtlen P, Losch-Beridon T, Mareya S, Schneider J. Capsule and Sprinkle Formulations of Lubiprostone Are Not Biologically Similar in Patients with Functional Constipation. Adv Ther. 2021 Jun;38(6):2936-2952. doi: 10.1007/s12325-021-01707-9. Epub 2021 Apr 8. PMID 33834354

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited in the United States
Pre-assignment Details: Treatment periods for Cohorts 1 and 2 did not have the same participants.
  Participants in each cohort were randomized to sequence.
  In each sequence the first treatment was given for 14 days, there was a 7-day washout period, and then the second treatment was given for 14 days.
Groups:
- Cohort 1: Treatment A Then Treatment B: Participants in Cohort 1 who received Treatment A: Lubiprostone Capsule, Fasted for 14 days, followed (after a 7-day washout) by Treatment B: Sprinkle Formulation, Fasted for 14 days
- Cohort 1: Treatment B Then Treatment A: Participants in Cohort 1 who received Treatment B: Sprinkle Formulation, Fasted for 14 days, followed (after a 7-day washout) by Treatment A: Lubiprostone Capsule, Fasted for 14 days
- Cohort 2: Treatment C Then Treatment D: Participants in Cohort 2 who received Treatment C: Sprinkle, Fed for 14 days, followed (after a 7-day washout) by Treatment D: Sprinkle Formulation, Fasted for 14 days
- Cohort 2: Treatment D Then Treatment C: Participants in Cohort 2 who received Treatment D: Sprinkle Formulation, Fasted for 14 days, followed (after a 7-day washout) by Treatment C: Sprinkle, Fed for 14 days
Period: Cohort 1
Arm/Group | Cohort 1: Treatment A Then Treatment B | Cohort 1: Treatment B Then Treatment A | Cohort 2: Treatment C Then Treatment D | Cohort 2: Treatment D Then Treatment C
Started (Participants in Cohort 2 were not included in the first treatment period) | 18 | 17 | 0 | 0
Completed | 14 | 17 | 0 | 0
Not Completed | 4 | 0 | 0 | 0
Period: Cohort 2
Arm/Group | Cohort 1: Treatment A Then Treatment B | Cohort 1: Treatment B Then Treatment A | Cohort 2: Treatment C Then Treatment D | Cohort 2: Treatment D Then Treatment C
Started (Participants from Cohort 1 were not included in the second treatment period) | 0 | 0 | 7 (New participants were enrolled for Cohort 2) | 7
Completed | 0 | 0 | 7 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population, defined as all randomized participants who took at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Treatment A Then Treatment B | Cohort 1: Treatment B Then Treatment A | Cohort 2: Treatment C Then Treatment D | Cohort 2: Treatment D Then Treatment C | Total
Number analyzed (Participants) | 18 | 17 | 7 | 7 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 17 | 7 | 7 | 49
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 4 | 4 | 27
  Male | 9 | 7 | 3 | 3 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 9 | 3 | 2 | 26
  Not Hispanic or Latino | 6 | 8 | 4 | 5 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 2 | 4 | 12
  White | 15 | 14 | 4 | 3 | 36
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 17 | 7 | 7 | 49

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1: Area Under the Concentration-time Curve (AUC) From Hour 0 to the Last Measurable Concentration (AUC0-t) of M3 Metabolite
Time Frame: 1 day
Population: PK population, defined as those with plasma concentration of lubiprostone or M3 sufficient to calculate at least 1 PK parameter
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Groups:
- Treatment A: Lubiprostone Capsule, Fasted: Participants in the pharmacokinetic-evaluable (PK) population who received treatment A
- Treatment B: Sprinkle Formulation, Fasted: Participants in the PK population who received treatment B
Arm/Group | Treatment A: Lubiprostone Capsule, Fasted | Treatment B: Sprinkle Formulation, Fasted
Number analyzed (Participants) | 31 | 31
h*pg/mL | 117.518 (57.56) | 163.615 (47.45)
Statistical Analysis 1: Comparison: Treatment A: Lubiprostone Capsule, Fasted vs Treatment B: Sprinkle Formulation, Fasted; Test type: Superiority; Ratio of Geometric LS Means = 1.441, 90% CI 2-sided [1.166 to 1.782]

2. Primary Outcome: Cohort 1: Maximum Observed Concentration (Cmax) of M3 Metabolite
Time Frame: 1 day
Population: Evaluable PK Population included all participants in the PK Population who had sufficient plasma drug concentration data of either lubiprostone or M3 to calculate at least 1 evaluable PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Groups:
- Treatment A: Lubiprostone Capsule, Fasted: Cohort 1 participants who received Treatment A
- Treatment B: Sprinkle Formulation, Fasted: Cohort 1 participants who received Treatment B
Arm/Group | Treatment A: Lubiprostone Capsule, Fasted | Treatment B: Sprinkle Formulation, Fasted
Number analyzed (Participants) | 31 | 31
pg/mL | 63.463 (55.56) | 127.729 (61.32)
Statistical Analysis 1: Comparison: Treatment A: Lubiprostone Capsule, Fasted vs Treatment B: Sprinkle Formulation, Fasted; Test type: Superiority; Ratio of Geometric LS Means = 2.045, 90% CI 2-sided [1.615 to 2.589]

3. Secondary Outcome: Cohort 2: Total Exposure (AUC0-t) of M3 With Administration of Sprinkle Lubiprostone Under Fed Versus (vs) Fasted Condition
Time Frame: 1 day
Population: PK Evaluable Population.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Groups:
- Treatment C: Sprinkle Formulation, Fed: Cohort 2 participants who received Treatment C
- Treatment D: Sprinkle Formulation, Fasted: Cohort 2 participants who received Treatment D
Arm/Group | Treatment C: Sprinkle Formulation, Fed | Treatment D: Sprinkle Formulation, Fasted
Number analyzed (Participants) | 14 | 14
h*pg/mL | 135.805 (58.17) | 152.900 (26.96)
Statistical Analysis 1: Comparison: Treatment C: Sprinkle Formulation, Fed vs Treatment D: Sprinkle Formulation, Fasted; Test type: Other; Ratio of Geometric LS Means = 0.888, 90% CI 2-sided [0.675 to 1.168]

4. Secondary Outcome: Cohort 2: Maximum Observed Concentration (Cmax) of M3 Metabolite in Fed vs Fasted Conditions
Time Frame: 1 day
Population: PK Evaluable Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Treatment C: Sprinkle Formulation, Fed | Treatment D: Sprinkle Formulation, Fasted
Number analyzed (Participants) | 14 | 14
pg/mL | 48.192 (30.52) | 116.815 (31.93)
Statistical Analysis 1: Comparison: Treatment C: Sprinkle Formulation, Fed vs Treatment D: Sprinkle Formulation, Fasted; Test type: Other; Ratio of Geometric LS Means = 0.413, 90% CI 2-sided [0.339 to 0.502]

5. Other Pre Specified Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An SAE is any untoward medical occurrence that results in death;is life-threatening;requires inpatient hospitalization or prolongation of present hospitalization;results in persistent or significant disability/incapacity;is a congenital anomaly/birth defect;or is a medically important event that may not be immediately life-threatening or result in death or hospitalization, but may jeopardize the participant or may require intervention to prevent one of other outcomes listed in definition above, or involves suspected transmission via a medicinal product of an infectious agent.
Time Frame: From the first dose of study drug up to 28 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: Lubiprostone Capsule, Fasted | Treatment B: Sprinkle Formulation, Fasted | Treatment C: Sprinkle Formulation, Fed | Treatment D: Sprinkle Formulation, Fasted
Number analyzed (Participants) | 31 | 35 | 14 | 14
Participants
  Adverse Events | 13 | 23 | 6 | 6
  Serious Adverse Events | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 28 days
Groups:
- Treatment A: All participants who received lubiprostone 2x24 μg capsule once orally.
- Treatment B: All participants who received lubiprostone 2x24 μg sprinkle formulation once orally.
- Treatment C: All participants who received lubiprostone 2x24 μg sprinkle formulation once orally under fed conditions.
- Treatment D: All participants who received lubiprostone 2x24 μg sprinkle formulation once orally under fasted conditions.
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/35 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/35 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 13/31 | 23/35 | 6/14 | 6/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=31) | Treatment B (N=35) | Treatment C (N=14) | Treatment D (N=14)
Nausea (Gastrointestinal disorders) | 5 | 10 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 10 | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 3 | 5 | 1 | 2
Eructation (Gastrointestinal disorders) | 2 | 3 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 4 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 4 | 5 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 7 | 0 | 2
Presyncope (Nervous system disorders) | 2 | 0 | 0 | 0
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 3 | 2 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0
Flushing (Vascular disorders) | 0 | 2 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 1

LIMITATIONS AND CAVEATS:
Because AUC0-∞ could only be determined in a limited number of participants, AUC0-t was used for primary comparisons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other